CLINICAL TRIAL: NCT02061098
Title: Effect of an Ellagitannin Rich Pomegranate Extract on Cardiovascular Risk Markers in Overweight Healthy Subjects. A Double-blind, Cross-over, Dose-response, Randomized, Placebo-controlled Trial (The POMEcardio Study)
Brief Title: Effect of a Pomegranate Extract on Cardiovascular Risk Markers in Overweight Healthy Subjects
Acronym: POMEcardio
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Universidad Católica San Antonio de Murcia (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Full Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CEBAS-CSIC-4
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Overweight
Keywords: Pomegranate; Cardiovascular; Urolithins; Microbiota; Polyphenols; Nutraceutical; Dietary supplement
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomegranate extract (Experimental): Crossover and dose-response: Both groups A and B will consume pomegranate extract and placebo. Both groups will also consume two doses of pomegranate extract and placebo.
  Group A will consume 1 daily capsule of pomegranate extract and group B will consume 1 daily capsule of placebo for 3 weeks. After a wash-out period of 3 weeks, group A will consume 1 daily capsule of placebo and group B will consume 1 daily capsule of pomegranate extract for 3 weeks. After a washout period of 3 weeks, group A will consume 4 daily capsules of pomegranate extract for 3 weeks and group B will consume 4 daily capsules of placebo for 3 weeks. After a washout period of 3 weeks, group A will consume 4 daily capsules of placebo for 3 weeks and group B will consume 4 daily capsules of pomegranate for 3 weeks.
  Interventions: Dietary Supplement: Pomegranate extract-first dose-Group A; Dietary Supplement: Pomegranate extract-first dose-Group B; Dietary Supplement: Pomegranate extract-second dose-Group A; Dietary Supplement: Pomegranate extract-second dose-Group B
- Placebo (Placebo Comparator): Crossover and dose-response: Both groups A and B will consume pomegranate extract and placebo. Both groups will also consume two doses of pomegranate extract and placebo.
  Group A will consume 1 daily capsule of pomegranate extract and group B will consume 1 daily capsule of placebo for 3 weeks. After a wash-out period of 3 weeks, group A will consume 1 daily capsule of placebo and group B will consume 1 daily capsule of pomegranate extract for 3 weeks. After a washout period of 3 weeks, group A will consume 4 daily capsules of pomegranate extract for 3 weeks and group B will consume 4 daily capsules of placebo for 3 weeks. After a washout period of 3 weeks, group A will consume 4 daily capsules of placebo for 3 weeks and group B will consume 4 daily capsules of pomegranate for 3 weeks.
  Interventions: Dietary Supplement: Placebo-first dose-Group B; Dietary Supplement: Placebo-first dose-Group A; Dietary Supplement: Placebo-second dose-Group B; Dietary Supplement: Placebo-second dose-Group A

INTERVENTIONS:
Dietary Supplement: Pomegranate extract-first dose-Group A — Group A will consume 1 daily capsule of pomegranate extract for 3 weeks
  Other Names: Group A consumes pomegranate extract (first dose)
  Arms: Pomegranate extract
Dietary Supplement: Placebo-first dose-Group B — Group B will consume 1 daily capsules of placebo for 3 weeks.
  Other Names: Group B consumes placebo (first dose)
  Arms: Placebo
Dietary Supplement: Pomegranate extract-first dose-Group B — After 3 weeks of washout, group B will consume 1 daily capsule of pomegranate extract for 3 weeks.
  Other Names: Group B consumes pomegranate extract (first dose)
  Arms: Pomegranate extract
Dietary Supplement: Placebo-first dose-Group A — After 3 weeks of washout, group A will consume 1 daily capsule of placebo for 3 weeks.
  Other Names: Group A consumes placebo (first dose)
  Arms: Placebo
Dietary Supplement: Pomegranate extract-second dose-Group A — After 3 weeks of washout, group A will consume 4 daily capsules of pomegranate extract for 3 weeks.
  Other Names: Group A consumes pomegranate extract (second dose)
  Arms: Pomegranate extract
Dietary Supplement: Placebo-second dose-Group B — After 3 weeks of washout, group B will consume 4 daily capsules of placebo for 3 weeks.
  Other Names: Group B consumes placebo (second dose)
  Arms: Placebo
Dietary Supplement: Pomegranate extract-second dose-Group B — After 3 weeks of washout, group B will consume 4 daily capsules of pomegranate extract for 3 weeks.
  Other Names: Group B consumes pomegranate extract (second dose)
  Arms: Pomegranate extract
Dietary Supplement: Placebo-second dose-Group A — After 3 weeks of washout, group A will consume 4 daily capsules of placebo for 3 weeks.
  Other Names: Group A consumes placebo (second dose)
  Arms: Placebo

SUMMARY:
The investigators objective is to carry out a placebo-controlled, dose-response, randomized clinical trial to assess the effects of polyphenols or derived metabolites on cardiovascular disease risk in overweight adult subjects upon the consumption of pomegranate extract.

The investigators hypothesis is that chronic consumption of a ellagitannin-rich source such as pomegranate extract could decrease serum oxidized-LDL as well as other inflammatory markers. The correlation between the effect exerted and the subjects' microbiota (capacity to produce the ellagitannin-derived metabolites urolithins) will indicate a possible role of urolithins on the effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-65 years
* Body mass index (BMI) >27 kg/m2
* Healthy status (no illness in the previous 3-months).

Exclusion Criteria:

* Smoking.
* Pregnancy/lactation.
* Severe medical illness/chronic disease/ or gastrointestinal pathology (ulcers, irritable bowel syndrome, ulcerative colitis, Crohn disease etc.).
* Previous gastrointestinal surgery
* Recent use of antibiotics (within 1-month prior to the study)
* Suspected hypersensitivity to pomegranate or any of its components
* Consumption of nutraceuticals, botanical extracts or other vitamin supplements or taking medication.
* Regular consumption of ellagitannin-containing foodstuffs (walnuts, pomegranate, strawberries, raspberries, oak-aged red wine) (after filling a food-frequency questionnaire).
* Intake of ellagitannins-containing foodstuffs the week before the pharmacokinetic intervention.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in serum oxidized LDL-cholesterol concentration | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  Effect on circulating levels of oxidized particles of LDL-cholesterol

SECONDARY OUTCOMES:
Change in serum lipids and lipoproteins levels | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  Effects on serum total cholesterol, LDL-cholesterol, HDL-cholesterol and apolipoproteins A1 (ApoA1), B (ApoB) and E (ApoE).
Change in serum sICAM, sVCAM and hsCRP | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  Effect on soluble intercellular adhesion molecule (sICAM), soluble vascular adhesion molecule (sVCAM) and high-sensitivity C-reactive protein (hsCRP)
Change in fecal microbiota | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  Prebiotic effect: Change in short fatty acids, bifidobacteria, lactobacilli and other selected species in feces
Number of volunteers with adverse events as a measure of safety and tolerability | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  * Change in markers involved in hepatic and renal functions: GGT, AST, ALP, ALT, CPK, urate, creatinin, albumin, bilirubin, LDH.
  * Change in hematological variables: leucocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, hemoglobin, hematocrit, mean corpuscular volume, mean platelet volume, platelets, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration.
  * Intolerance, dyspepsia, allergic reactions, constipation, diarrhea, abdominal pain, nausea.
Change in phenolics and derived metabolites in plasma, feces and urine. | Change from baseline at 3, 6, 9, 12, 15, 18, 21 and 24 weeks
  Dose-response effect of pomegranate intake on phenolics and gut-microbiota derived metabolites in plasma, feces and urine.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Juan Carlos Espín, PhD, Principal Investigator — National Research Council (CEBAS-CSIC, Murcia, Spain)
Locations (1):
- UCAM (San Antonio Catholic University from Murcia), Murcia, Murcia, Spain